CLINICAL TRIAL: NCT01769170
Title: A Phase 3 Study of the Safety, Tolerability, and Efficacy of CMX001 for the Prevention of Cytomegalovirus (CMV) Infection in CMV-seropositive (R+) Hematopoietic Stem Cell Transplant Recipients
Brief Title: A Study of the Safety and Efficacy of CMX001 for the Prevention of CMV Infection in CMV-seropositive HCT Recipients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CMX001-301
Record Dates: First submitted 2013-01-14; First posted 2013-01-16 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: CMV
Keywords: CMV; Hematopoietic Stem Cell Transplant Recipients; Prevention
MeSH Terms: interventions — brincidofovir

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Matching placebo administered orally twice weekly
  Interventions: Other: Placebo
- Brincidofovir (Active Comparator): 100 mg brincidofovir administered orally twice weekly
  Interventions: Drug: Brincidofovir

INTERVENTIONS:
Drug: Brincidofovir
  Other Names: BCV; CMX001; Hexadecyloxypropyl cidofovir; HDP-CDV
  Arms: Brincidofovir
Other: Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel group, multicenter study compared the effectiveness of oral brincidofovir (BCV) to placebo for the prevention of cytomegalovirus (CMV) infection in stem cell transplant patients who were CMV seropositive but negative for CMV viremia before starting treatment with BCV.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, parallel group multicenter study of oral brincidofovir (BCV) in approximately 450 cytomegalovirus (CMV)-seropositive subjects who had undergone allogeneic hematopoietic stem cell transplantation (HCT). The study consisted of a screening evaluation and a treatment phase of 10 to 14 weeks. Dosing with the study drug (BCV or placebo) was initiated as soon as individual subjects could ingest tablets after transplant but no later than Day 28 post-transplant, and was continued through Week 14. All randomized subjects remained on study and followed the same scheduled study treatment. Study assessments were performed weekly from randomization through completion of the first post-treatment follow-up assessment at Week 15, and every 3 weeks thereafter through Week 24.

ELIGIBILITY:
Inclusion Criteria

Subjects were required to meet all of the following criteria, as applicable, to be eligible to participate in this study:

1. Were allogeneic hematopoietic stem cell transplant (HCT) recipients who had prior evidence of cytomegalovirus (CMV) exposure (CMV-seropositive) before transplantation and were CMV viremia negative at screening and at any other assessments performed prior to the first dose of study drug.
2. Were aged ≥18 years.
3. If male, were willing to use an acceptable contraceptive method(s) throughout the duration of his participation in the study, i.e., through Week 24, when engaging in sexual intercourse with a female subject of childbearing potential.
4. If female of childbearing potential, i.e., not postmenopausal or surgically sterile, were willing to use 2 acceptable contraceptive methods, 1 of which must have been a barrier method, throughout the duration of her participation in the study, i.e., through Week 24, when engaging in sexual intercourse with a nonsterile male partner.
5. Were able to begin study drug dosing within 28 days following the qualifying HCT.
6. Were able to comfortably ingest and absorb oral medication (in the judgment of the investigator and base don lack of significant gastrointestinal events/medical history).
7. Were willing and able to understand and provide written informed consent.
8. Were willing and able to participate in all required study activities for the entire duration of the study (i.e., through Week 24).

Exclusion Criteria

Subjects who met any of the following criteria, as applicable, were not eligible to participate in this study:

1. Was pregnant or planned to become pregnant during the anticipated duration of her participation in the study (i.e., through Week 24), or was nursing a child.
2. Had a positive CMV viremia test (at the designated central virology laboratory or a local virology laboratory) at any time between transplant and the first dose of study drug.
3. Weighed ≥120 kg (~265 lbs).
4. Had hypersensitivity (not renal dysfunction or eye disorder) to cidofovir (CDV), brincidofovir (BCV), or its excipients.
5. Had received (or were anticipated to need treatment with) any of the following:

   * Ganciclovir, valganciclovir, foscarnet, intravenous CDV, or any other anti-CMV therapy (including CMV immune globulin, cell-based therapies, and investigational anti-CMV drugs, e.g., leflunomide, letermovir, or maribavir) at any time post-transplant;
   * Any anti-CMV vaccine at any time;
   * Any other investigation drug within 14 days prior to the first dose of study drug (unless prior approval had been received from the Chimerix medical monitor or designee); or
   * Prior treatment with BCV at any time.
6. Were receiving of the following drugs on the first dose of study drug or were anticipated to receive any of these drugs at the doses described after the first dose of study drug:

   * Acyclovir orally at >2000 mg total daily dose (TDD) or intravenously at >15 mg/kg TDD;
   * Valaciclovir at >3000 mg TDD; or
   * Leflunomide at any dose.
7. Were receiving digoxin or ketoconazole (other than topical formulations) at the first dose of study drug or were anticipated to need treatment with either digoxin or ketoconazole during the treatment phase (through Week 14).
8. Had possible, probably, or definitive CMV disease diagnosed within 6 months prior to first dose of study drug.
9. Were infected with HIV (based on serology), or had an active hepatitis C virus (HCV) or hepatitis B virus (HBV) infection, as evidence by detectable plasma HCV RNA or HBV DNA, respectively.
10. Had received another allogeneic HCT (i.e., other than the qualifying HCT) within 2 years prior to the first dose of study drug.
11. Had renal insufficiency, as evidence by an estimated glomerular filtration rate (eGFR) <15 mL/min or required renal dialysis.
12. Had hepatic abnormalities as evidence by a screening of alanine aminotransferase or aspartate aminotransferase >5 x the upper limit of normal (ULN), as reported by the central safety laboratory.
13. Had a screening total bilirubin >2 x the ULN and direct bilirubin >1.5 x the ULN, as reported by the central safety laboratory.
14. Had active solid tumor malignancies with the exception of basal cell carcinoma or the underlying condition necessitating HCT (e.g., lymphomas).
15. Had Stage 2 or higher graft versus host disease of the gut or any other GI disease that would have, in the judgment of the investigator, precluded the subject from taking or absorbing oral medication (e.g., clinically active Crohn's disease, ischemic colitis, moderate or severe ulcerative colitis, small bowel resection, ileus, or any condition expected to require abdominal surgery during the course of study participation).
16. Had any other condition, including abnormal laboratory values, that would have, in the judgement of the investigator, put the subject at increased risk by participating in the study or would have interfered with the conduct or planned analyses of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 452 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (39):
  - University of California, San Diego-Moores Cancer Center, La Jolla, California
  - UCLA Medical Center, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Colorado Blood Cancer Institute, Denver, Colorado
  - University of Miami Hospital, Miami, Florida
  - Winship Cancer Institute-Emory, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - The Universit of Iowa, Iowa City, Iowa
  - Johns Hopkins University, Baltimore, Maryland
  - Beth Isreal Decaconess Medical Center, Boston, Massachusetts
  - Brigham and Womens Hospital, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Harper University Hospital, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Hackensack University, Hackensack, New Jersey
  - Mt. Sinai Medical Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Weill Cornell Medical College/NY Presbyterial Hospital, New York, New York
  - Montefiore Medical Center, The Bronx, New York
  - Levine Cancer Institute/Carolinas Health, Charlotte, North Carolina
  - Duke Cancer Institute, Durham, North Carolina
  - Wake Forest, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - The Jewish Hospital, Cincinnati, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny-Singer Research Institute, Pittsburgh, Pennsylvania
  - Western Pennsylvania Hospital, Pittsburgh, Pennsylvania
  - Hollings Cancer Center, Charleston, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Methodist Healthcare of San Antonio, San Antonio, Texas
  - University of Utah, Huntsman Cancer Institute, Salt Lake City, Utah
  - Intermountain Healthcare, Salt Lake City, Utah
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
- Belgium (2):
  - Centre Hospitalier Universitaire Sart Tilman Liege, Brussels, Liege
  - Cliniques Universitaires Saint Luc, Brussels
- Canada (2):
  - University of Toronto, Toronto, Ontario
  - Centre Hospitalier Universitaire de Montreal, Hopital Maisonneuve-Rosemont, Montreal, Quebec

REFERENCES:
- [Result] Marty FM, Winston DJ, Chemaly RF, Mullane KM, Shore TB, Papanicolaou GA, Chittick G, Brundage TM, Wilson C, Morrison ME, Foster SA, Nichols WG, Boeckh MJ; SUPPRESS Trial Clinical Study Group. A Randomized, Double-Blind, Placebo-Controlled Phase 3 Trial of Oral Brincidofovir for Cytomegalovirus Prophylaxis in Allogeneic Hematopoietic Cell Transplantation. Biol Blood Marrow Transplant. 2019 Feb;25(2):369-381. doi: 10.1016/j.bbmt.2018.09.038. Epub 2018 Oct 4. PMID 30292744

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Brincidofovir | Placebo
Started | 303 | 149
Completed | 232 | 122
Not Completed | 71 | 27

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat Analysis Set, which included all randomized subjects who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brincidofovir | Placebo | Total
Number analyzed (Participants) | 303 | 149 | 452
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (14.29) | 51.9 (15.03) | 52.6 (14.53)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163 | 98 | 261
  Male | 140 | 51 | 191

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Clinically Significant CMV Infection Through Week 24 Post-Transplant
Description: Clinically significant cytomegalovirus (CMV) infection was defined by either of the following outcomes:
  1. Onset of CMV end-organ disease; or
  2. Initiation of anti-CMV-specific preemptive therapy based on documented CMV viremia (as measured by the central virology laboratory) and the clinical condition of the subject.
  CMV viremia (i.e., the measurement of CMV DNA in plasma) was determined by the designated central virology laboratory at all scheduled visits via quantitative polymerase chain reaction (qPCR) testing using the Roche COBAS® AmpliPrep/COBAS® TaqMan® CMV Test.
Time Frame: 24 weeks
Population: Intent-to-Treat Analysis Set, which included all subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Brincidofovir | Placebo
Number analyzed (Participants) | 303 | 149
Participants | 155 | 78

2. Secondary Outcome: Incidence of Clinically Significant CMV Infection Through Week 14
Description: The incidence of clinically significant cytomegalovirus (CMV) infection through Week 14.
  Blood and urine for virologic evaluations were collected at screening, pre-dose on the first day of study drug administration, and at pre-specified intervals throughout the treatment phases of the study and sent to a designated central virology laboratory for analysis. Blood samples were used for real-time assay of CMV viremia in plasma using a qPCR assay. Urine samples were stored for possible future retrospective analyses of CMV.
Time Frame: 14 weeks
Population: Intention-to-Treat Analysis Set, which included all randomized subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Brincidofovir | Placebo
Number analyzed (Participants) | 303 | 149
Participants | 74 | 57

ADVERSE EVENTS:
Arm/Group | Brincidofovir | Placebo
Serious Adverse Events (participants affected / at risk) | 173/303 | 56/149
Other Adverse Events (participants affected / at risk) | 302/303 | 146/149
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Brincidofovir (N=303) | Placebo (N=149)
Acute graft versus host disease (Immune system disorders) | 98 | 9
Chronic graft versus host disease (Immune system disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 9 | 0
Pneumonia (Infections and infestations) | 5 | 4
Cellulitis (Infections and infestations) | 3 | 1
BK virus infection (Infections and infestations) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 2 | 0
Corona virus infection (Infections and infestations) | 2 | 0
Enterovirus infection (Infections and infestations) | 1 | 1
Metapneumovirus infection (Infections and infestations) | 1 | 1
Rhinovirus infection (Infections and infestations) | 1 | 1
Sepsis (Infections and infestations) | 1 | 1
Septic shock (Infections and infestations) | 2 | 0
Staphylococcal infection (Infections and infestations) | 0 | 2
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Toxoplasmosis (Infections and infestations) | 2 | 0
Adenovirus infection (Infections and infestations) | 1 | 0
Bacterial infection (Infections and infestations) | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0
Cystitis viral (Infections and infestations) | 0 | 1
Cystitis klebsiella (Infections and infestations) | 1 | 0
Encephalitis (Infections and infestations) | 0 | 1
Enterococcal sepsis (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Gastroenteritis norovirus (Infections and infestations) | 1 | 0
Gastroenteritis rotavirus (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 0 | 1
Human herpesvirus 6 infection (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 1 | 0
Nocardiosis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Pneumonia haemophilus (Infections and infestations) | 0 | 1
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia parainfluenza viral (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 1 | 0
Pneumonia viral (Infections and infestations) | 1 | 0
Respiratory syncytial virus infection (Infections and infestations) | 1 | 0
Rotavirus infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Systemic candida (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Viral haemorrhagic cystitis (Infections and infestations) | 1 | 0
Zygomycosis (Infections and infestations) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 4
Nausea (Gastrointestinal disorders) | 5 | 1
Abdominal pain (Gastrointestinal disorders) | 5 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Enteritis (Gastrointestinal disorders) | 2 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Colonic pseudo-obstruction (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileal perforation (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Pneumatosis intestinalis (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 9 | 8
Multi-organ failure (General disorders) | 4 | 1
Chest pain (General disorders) | 1 | 0
Drug withdrawal syndrome (General disorders) | 1 | 0
Gait disturbance (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 1
Aspartate aminotransferase increased (Investigations) | 4 | 1
Klebsiella test positive (Investigations) | 2 | 1
Polyomavirus test positive (Investigations) | 2 | 1
Bacterial test positive (Investigations) | 0 | 2
Escherichia test positive (Investigations) | 1 | 1
Staphylococcus test positive (Investigations) | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1
Citrobacter test positive (Investigations) | 0 | 1
Electrocardiogram Qt prolonged (Investigations) | 1 | 0
Enterococcus test positive (Investigations) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Human rhinovirus test positive (Investigations) | 1 | 0
Pseudomonas test positive (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diffuse alveolar damage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute myeloid leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 6 | 3
Leukaemia recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Burkitt's lymphoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasma cell leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 5 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hypophagia (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 9 | 4
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal tubular necrosis (Renal and urinary disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0
Jugular vein thrombosis (Vascular disorders) | 2 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Microangiopathic haemolytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 4 | 0
Supraventricular tachycardia (Cardiac disorders) | 3 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Intracardiac thrombus (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 4 | 1
Transplant failure (Injury, poisoning and procedural complications) | 2 | 2
Delayed engraftment (Injury, poisoning and procedural complications) | 1 | 1
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Syncope (Nervous system disorders) | 2 | 1
Seizure (Nervous system disorders) | 1 | 1
Arachnoiditis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 4 | 0
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Venoocclusive liver disease (Hepatobiliary disorders) | 2 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0
Hepatitis acute (Hepatobiliary disorders) | 1 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Brincidofovir (N=303) | Placebo (N=149)
Diarrhoea (Gastrointestinal disorders) | 184 | 54
Abdominal pain (Gastrointestinal disorders) | 104 | 26
Nausea (Gastrointestinal disorders) | 93 | 29
Vomiting (Gastrointestinal disorders) | 74 | 25
Constipation (Gastrointestinal disorders) | 29 | 11
Dry mouth (Gastrointestinal disorders) | 21 | 13
Abdominal distension (Gastrointestinal disorders) | 19 | 10
Dyspepsia (Gastrointestinal disorders) | 24 | 4
Decreased appetite (Metabolism and nutrition disorders) | 67 | 19
Hyperglycaemia (Metabolism and nutrition disorders) | 48 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 47 | 10
Hypomagnesaemia (Metabolism and nutrition disorders) | 38 | 12
Hyponatraemia (Metabolism and nutrition disorders) | 21 | 8
Hyperkalaemia (Metabolism and nutrition disorders) | 20 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 21 | 5
Dehydration (Metabolism and nutrition disorders) | 20 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 19 | 4
Hypophosphataemia (Metabolism and nutrition disorders) | 17 | 4
Fatigue (General disorders) | 42 | 28
Oedema peripheral (General disorders) | 52 | 18
Pyrexia (General disorders) | 42 | 27
Mucosal inflammation (General disorders) | 32 | 15
Asthenia (General disorders) | 29 | 6
Acute graft versus host disease (Immune system disorders) | 173 | 48
Hypogammaglobulinaemia (Immune system disorders) | 16 | 6
BK virus infection (Infections and infestations) | 24 | 7
Clostridium difficile colitis (Infections and infestations) | 27 | 3
Cystitis viral (Infections and infestations) | 17 | 4
Alanine aminotransferase increased (Investigations) | 34 | 9
Aspartate aminotransferase increased (Investigations) | 29 | 8
Blood creatinine increased (Investigations) | 24 | 12
Weight decreased (Investigations) | 24 | 2
Rash (Skin and subcutaneous tissue disorders) | 43 | 28
Pruritus (Skin and subcutaneous tissue disorders) | 29 | 13
Dry skin (Skin and subcutaneous tissue disorders) | 27 | 8
Erythema (Skin and subcutaneous tissue disorders) | 16 | 4
Headache (Nervous system disorders) | 31 | 21
Dizziness (Nervous system disorders) | 22 | 13
Tremor (Nervous system disorders) | 20 | 10
Dysgeusia (Nervous system disorders) | 18 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 31 | 20
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 20 | 7
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 15 | 9
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 10 | 8
Pain in extremity (Musculoskeletal and connective tissue disorders) | 26 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 22 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 13 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 8
Acute kidney injury (Renal and urinary disorders) | 30 | 10
Pollakiuria (Renal and urinary disorders) | 20 | 10
Dysuria (Renal and urinary disorders) | 17 | 10
Insomnia (Psychiatric disorders) | 31 | 12
Depression (Psychiatric disorders) | 20 | 6
Anxiety (Psychiatric disorders) | 14 | 10
Hypertension (Vascular disorders) | 33 | 16
Hypotension (Vascular disorders) | 32 | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 19 | 11
Anaemia (Blood and lymphatic system disorders) | 18 | 7
Neutropenia (Blood and lymphatic system disorders) | 16 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 16 | 3
Dry eye (Eye disorders) | 15 | 11
Tachycardia (Cardiac disorders) | 18 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Within 12 months after the end of the Study at all sites, if no publication of the overall multi-center results has been made, institutions are entitled to publish their locally obtained results, provided the Sponsor is given opportunity to review and comment. Institution publications may be delayed up to an additional 60 days to allow Sponsor to seek patent protection.